CLINICAL TRIAL: NCT05018910
Title: Investigating the Impact of Skin to Skin on Preterm Infant Heart Rate Variability
Brief Title: Skin to Skin and Heart Rate Variability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Jessie R. Maxwell, Assistant Professor of Pediatrics and Neurosciences, University of New Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ID: 21-177
Record Dates: First submitted 2021-08-17; First posted 2021-08-24 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-09

CONDITIONS: Heart Rate Variability; Preterm Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: All infants enrolled in the study had their heart rate variability measured before, during, and after skin-to-skin sessions. There was no randomization or testing of efficacy.
Masking Description: All infants enrolled had their heart rate variability measured.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heart Rate Variability (Other): All infants enrolled in the study had their heart rate variability measured before, during, and after skin-to-skin sessions. This was the only arm of the study.
  Interventions: Other: Skin to Skin

INTERVENTIONS:
Other: Skin to Skin — During routine Skin-to-skin sessions, the heart rate variability of the infant will be measured.

SUMMARY:
The objective of this study is to monitor heart rate variability in preterm infants receiving respiratory support, including conventional mechanical ventilation, during skin-to-skin care. We hypothesize that skin to skin care will be associated with a more mature pattern of parasympathetic activity as measured by various domains of heart rate variability. Specifically, the standard deviation of the normal-to-normal interval (SDNN), the root mean squared of successive differences of normal-to-normal intervals (RMSDD), and the standard deviation of deceleration (SDDec) will decrease in infants that are receiving skin-to-skin care across all types of respiratory support compared to infants who are lying in their isolette.

DETAILED DESCRIPTION:
This will be a prospective crossover study, with each infant serving as their own control. Any infant for whom the parent has consented to participate in the study will have heart rate variability leads applied and be monitored before, during and after a skin-to-skin session with the infant's parent. Due to the nature of the study, blinding is not feasible. Infants will remain on the hospital cardiac monitor during the study to maintain standard of care, and data obtained in this study will not be used for clinical care. All sessions will occur during the infant's NICU admission.

Infants will be screened for eligibility by reviewing the Newborn Intensive Care Unit (NICU) census daily. Consent will be obtained after an infant has delivered. No pregnant women will be approached for consent.

Any infant who has been consented for participation and completes at least 1 skin to skin session will be included in the final study sample. As skin to skin is part of standard of care, and information, aside from gender, will not be obtained from the parent, consent will be obtained for the infant to participate in the study.

This study is observational because there was no randomization (no intervention).

ELIGIBILITY:
Inclusion Criteria:

* Infants must be less than or equal to 30 weeks gestational age at time of delivery.
* Both inborn and outborn infants are eligible for this study.
* Infants must be less than 6 weeks postnatal age.
* Infants must have had a cranial ultrasound with results showing no intraventricular severe intraventricular hemorrhage (Grade III or IV) [10].
* Infants must require respiratory support at the time of the first session. This will include mechanical ventilation, noninvasive positive pressure ventilation (NIPPV), continuous positive airway pressure (CPAP), high flow nasal cannula (HFNC) or low flow nasal cannula (LFNC).
* Consenting biological or legal adoptive mother of the infant must speak English. If the study is unable to enroll an appropriate number of patients, will consider including non-English speaking patients. However, due to limited resources for this study, we will start with only English-speaking patients. Biological or legal adoptive mother will provide consent for the infant to participate in this study.
* Biological or legal adoptive fathers of the infant are eligible to complete skin to skin sessions with the infant. As we are not collecting any information from the father, and skin to skin is a part of accepted standard of care, consent will not be obtained from the father.
* Infants of employees are eligible to participate. Undue influence or coercion will not be applied to infants of employees and participation or lack thereof will not affect employment status.

Exclusion Criteria:

* Infants who have not received a head ultrasound.
* Infants with grade III or higher intraventricular hemorrhage identified on a head ultrasound.
* Infants on high frequency ventilation, due to the artifact transmitted to ECG.
* Infants with known genetic disorders or known prenatal chromosomal anomalies.
* Infants with one or more major congenital anomaly.
* Infants undergoing active sepsis evaluation or treatment for infection.
* Infants on blood pressure or cardiac medications or infusions including inotropic mediations.
* Mothers (biological or legal adoptive) that are <18 years of age will not be approached for consent.
* Mothers (biological or legal adoptive) who are unable to provide consent due to having a legal representative will not be approached for consent in this study.
* Mothers (biological or legal adoptive) who are prisoners will not be approached for this study as participation requires multiple skin to skin session with the infant

Ages: 1 Day to 6 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2021-07-04 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- HRV Monitoring: All infants consented for the study had heart rate variability monitored before, during and after a skin-to-skin with the caregiver. All infants had the heart rate variability completed; infants were not treated differently. If an infant was consented for the study, the heart rate variability was recorded during an already planned skin-to-skin session with the caregiver.
  The "before period" of the skin-to-skin session was NO skin-to-skin heart rate variability (pre); during skin to skin was heart rate variability during the session; the after period of the skin-to-skin session was NO skin-to-skin heart rate variability (post) but obtained after the session.
Period: Overall Study
Arm/Group | HRV Monitoring
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- HRV Monitoring: All infants consented for the study had heart rate variability monitored before, during and after a skin-to-skin with the caregiver.
Arm/Group | HRV Monitoring
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: gestational age in weeks] | 29 [25.5 to 29.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  United States | 10
Respiratory support during Heart rate variability (HRV) [Number; unit: type of respiratory support]
  Continuous positive pressure | 7
  Nasal canula | 3

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate Variability
Description: The standard deviation of the normal-to-normal interval, the root mean squared of successive differences of normal-to-normal intervals and the standard deviation of deceleration will be measured before, during and after a skin to skin sessions.
Time Frame: up to 2 hours duration
Measure: Median (Inter-Quartile Range); unit: ms
Groups:
- HRV Monitoring: All infants consented for the study had heart rate variability monitored before, during and after a skin-to-skin with the caregiver.
  The outcome measure provided is the Standard Deviation of the normal-to-normal interval (SDNN) obtained after the session was completed.
Arm/Group | HRV Monitoring
Number analyzed (Participants) | 10
ms | 9.68 [1.45 to 17.91]

ADVERSE EVENTS:
Time Frame: Duration of enrollment (1.5 years)
Groups:
- HRV Monitoring: All infants consented for the study had heart rate variability monitored before, during and after a skin-to-skin with the caregiver. There were not separate groups.
Arm/Group | HRV Monitoring
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-21): https://cdn.clinicaltrials.gov/large-docs/10/NCT05018910/Prot_SAP_000.pdf